CLINICAL TRIAL: NCT06072235
Title: Facemasks and COVID-19 Pandemic in Chronic Pain Patients With Hearing Impairment
Brief Title: Facemasks and Chronic Pain Patients With Hearing Loss
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Salem2018 HearLoss Pain Mask
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hearing Loss; Chronic Pain
MeSH Terms: conditions — Hearing Loss; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Verbal communication — Verbal communication; by talking and listening

SUMMARY:
Facemasks may impede communication. Impaired communication may worsen healthcare outcomes. This study explores the problem of hearing impairment in chronic pain patients, and the impact of facemasks on healthcare outcomes in chronic pain patients.

Data collection includes patient's age, anxiety score, depression score, numeric pain score, and effects of facemasks on treatment outcomes. Pain is measured using numeric pain rating scale. Depression is measured using the Patient Health Questionnaire (PHQ-9) scale. Anxiety is measured using the General Anxiety Disorder (GAD-7) scale.

DETAILED DESCRIPTION:
Facemasks may impede communication. Impaired communication may worsen healthcare outcomes. There is inadequate data on the prevalence of hearing impairment in chronic pain patients. There is inadequate information about the impact of facemasks on treatment outcomes in chronic pain patients with hearing impairment. This prospective study explores the problem of hearing impairment in chronic pain patients, and the impact of facemasks on healthcare outcomes in chronic pain patients.

This is a prospective cohort study of adult patients undergoing pain treatment at an interventional pain clinic in Canada. Data collection includes patient's age, anxiety score, depression score, analgesic usage, numeric pain score, and effects of facemasks on pain management outcomes. Pain is measured using numeric pain rating scale of 0-10, with change of 2-points being considered significant. Depression is measured using the Patient Health Questionnaire (PHQ-9) scale of 0-27, with change of 3-points being considered significant. Anxiety is measured using the General Anxiety Disorder (GAD-7) scale of 0-21, with change of 3-points being considered significant.

Data are analyzed with IBM® SPSS® Statistics 25; using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adults
* chronic pain diagnosis
* diagnosed hearing impairment
* use of hearing aid

Exclusion Criteria:

* complete deafness
* cochlear implant
* severe vision impairment
* cognitive dysfunction

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of consecutive adult patients who underwent pain management at a pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Numeric pain score, objective measurement using validated Numeric Pain Rating scale | 12 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

SECONDARY OUTCOMES:
Depression score, objective measurement using validated Patient Health Questionnaire (PHQ-9) scale | 12 weeks
  Depression score, using the Patient Health Questionnaire (PHQ-9) scale of 0-27; low scores indicate less depression, high scores indicate worse depression
Anxiety score, objective measurement using validated General Anxiety Disorder (GAD-7) scale | 12 weeks
  Anxiety score, using the General Anxiety Disorder (GAD-7) scale of 0-21; low scores indicate less anxiety, high scores indicate worse anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No